CLINICAL TRIAL: NCT02441114
Title: A Pilot Study to Investigate Pharmacokinetic Characteristics After Co-administration of HCP0910 and HGP1011
Brief Title: Pharmacokinetics of Co-administration of Seretide 250 Diskus (HCP0910) and Spiriva Capsule for Inhalation (HGP1011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Clinical pharmacology and therapeutics, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HM_COPD_PILOT
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhalation of HCP0910 and HGP1011 (Experimental): Single, twice and triple inhalation of HCP0910 and HGP1011 (open-label, single-arm, dose-escalation) at period 1, 2, and 3, respectively.
  The periods were separated with a washout period of 14 days.
  Interventions: Drug: HCP0910 and HGP1011

INTERVENTIONS:
Drug: HCP0910 and HGP1011 — Inhalation of HCP0910 (Seretide 250 diskus (Fluticasone Propionate 250 mcg/Salmeterol Xinafoate 72.5 mcg)) and HGP1011 (Spiriva capsule for inhalation (Micronized Tiotropium Bromide Monohydrate 22.5 mcg))
  Other Names: Seretide 250 diskus and Spiriva capsule for inhalation; Fluticasone/Salmeterol and Tiotropium

SUMMARY:
This pilot study was designed to evaluate the pharmacokinetic characteristics of fluticasone, salmeterol, and tiotropium after co-administration of HCP 0910 (Seretide 250 diskus) and HGP1011 (Spiriva capsule for inhalation) which are prescribed concomitantly for the patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Within 3 weeks prior to the first administration of study drug, volunteers who agreed the participation of this study by their written consent will undergo screening, including physical examination and clinical laboratory test etc, to evaluate whether they are eligible to participate in this study. Study drugs will be administered at about 8 A.M. in the morning of the drug administration day, followed by blood collection for evaluation of pharmacokinetics. The same schedule with increased dose will be proceeded after 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects (at screening)
* Body weight between 55kg - 90kg, BMI (Body Mass Index) between 18.0 - 27.0
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent

Exclusion Criteria:

* Volunteer who has past or present history of any diseases such as liver including hepatitis virus carrier, kidney, Neurology, immunology, pulmonary, endocrine, hematooncology, cardiology, mental disorder
* Volunteer who had drug(Aspirin, antibiotics) hypersensitivity reaction
* Subject who already participated in other trials in 3 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 months or transfusion

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period1
Arm/Group | Inhalation of HCP0910 and HGP1011
Started | 10
Completed | 10
Not Completed | 0
Period: Washout1
Arm/Group | Inhalation of HCP0910 and HGP1011
Started | 10
Completed | 10
Not Completed | 0
Period: Period2
Arm/Group | Inhalation of HCP0910 and HGP1011
Started | 10
Completed | 10
Not Completed | 0
Period: Washout2
Arm/Group | Inhalation of HCP0910 and HGP1011
Started | 10
Completed | 6
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Period3
Arm/Group | Inhalation of HCP0910 and HGP1011
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inhalation of HCP0910 and HGP1011
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (4.9)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUClast)
Description: Area under the concentration of fluticasone versus time curve from the time of dosing to the last measurable concentration
Time Frame: Period 1 (day 1), 2 (day 15), and 3 (day 29) at 0 to 24 h post-dose
Population: 10 subjects for period 1 and 2; 6 subjects for period 3
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Inhalation of HCP0910 and HGP1011
Number analyzed (Participants) | 10
h*pg/mL
  Period 1 | 686.98 (111.36)
  Period 2 | 1247.63 (276.51)
  Period 3 | 1769.58 (370.80)

2. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Time to maximum concentration of fluticasone
Time Frame: Period 1 (day 1), 2 (day 15), and 3 (day 29) at 0 to 24 h post-dose
Population: 10 subjects for period 1 and 2; 6 subjects for period 3
Measure: Median (Full Range); unit: h
Arm/Group | Inhalation of HCP0910 and HGP1011
Number analyzed (Participants) | 10
h
  Period 1 | 0.76 [0.33 to 3.00]
  Period 2 | 0.50 [0.08 to 1.50]
  Period 3 | 0.88 [0.33 to 1.50]

3. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration of fluticasone
Time Frame: Period 1 (day 1), 2 (day 15), and 3 (day 29) at 0 to 24 h post-dose
Population: 10 subjects for period 1 and 2; 6 subjects for period 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Inhalation of HCP0910 and HGP1011
Number analyzed (Participants) | 10
pg/mL
  Period 1 | 95.70 (20.14)
  Period 2 | 173.56 (44.32)
  Period 3 | 246.77 (57.30)

ADVERSE EVENTS:
Groups:
- HCP0910 and HGP1011: Single Inhalation of HCP0910 and HGP1011 (Open-label, Single-arm, Single dosing, Dose-escalation)
  HCP0910 and HGP1011: Inhalation of HCP0910 (Seretide 250 diskus (Fluticasone Propionate 250 mcg/Salmeterol Xinafoate 72.5 mcg)) and HGP1011 (Spiriva capsule for inhalation (Micronized Tiotropium Bromide Monohydrate 22.5 mcg))
Arm/Group | HCP0910 and HGP1011
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCP0910 and HGP1011 (N=10)
Diarrhoea (Gastrointestinal disorders) | 10 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No